CLINICAL TRIAL: NCT00503230
Title: Reducing Ethnic Health Disparities: Motivating HIV+ Latinos to Quit Smoking
Acronym: AURORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA018079 (NIH); R01DA018079 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Tobacco Dependence; HIV Infections
Keywords: tobacco; smoking; HIV; Latino
MeSH Terms: conditions — Tobacco Use Disorder; HIV Infections; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care Intervention (SCI) (Active Comparator)
  Interventions: Behavioral: Standard Care Intervention (SCI)
- Culturally Tailored Intervention (CTI) (Active Comparator)
  Interventions: Behavioral: Culturally Tailored Intervention (CTI)

INTERVENTIONS:
Behavioral: Standard Care Intervention (SCI) — Standard Care Intervention (SCI)
  Arms: Standard Care Intervention (SCI)
Behavioral: Culturally Tailored Intervention (CTI) — Culturally Tailored Intervention (CTI)
  Arms: Culturally Tailored Intervention (CTI)

SUMMARY:
The purpose of this study is to develop and evaluate a brief clinic-based culturally tailored smoking cessation treatment for a largely low-income, Latino, HIV+ population. We will compare this Culturally-Tailored Intervention (CTI) that incorporates a strong social support component and is targeted to the special needs and concerns of a Latino population to a Standard Care Intervention (SCI) control condition, in a randomized controlled trial. We hypothesize that those Latinos receiving the CTI will demonstrate greater biochemically verified smoking abstinence rates at 12-months post-baseline than those receiving the SCI control treatment. All study participants and their participating social supports will be offered use of the nicotine patch.

DETAILED DESCRIPTION:
Advances in the treatment of HIV-disease have shown dramatic effects on improving immune function in a significant proportion of people infected with HIV in the United States. For the first time since the beginning of the HIV epidemic, individuals with HIV are faced with the prospect of living longer, healthier lives. Cigarette smoking is highly prevalent among HIV+ individuals and, in addition to the negative health consequences commonly resulting from smoking, poses unique health risks to those with HIV. Our present research investigation, Positive PATHS (PATHS), the only NIH-funded smoking cessation study in HIV+ persons, is designed to evaluate a clinic-based motivational smoking cessation intervention among HIV+ smokers in Southern New England. Preliminary analysis of the PATHS investigation indicate that both a standard care intervention (brief advice and NRT) and a more extensive motivational counseling condition have similar biochemically verified smoking abstinence rates 6-months post intervention, with Latino participants responding better to the brief standard care condition. The goal of the current application is to expand upon the preliminary results of this study and target the standard care intervention to Latino HIV+ patients who were found to respond best to a brief directive approach. This expanded standard care approach will incorporate the use of culturally specific materials to provide brief advice to both the patient and a patient-identified social support person who will be trained in ways to support cessation efforts. Latinos are a population greatly affected by HIV and tobacco use, yet rarely discussed in existing research. Most tobacco research that includes Latinos has focused on prevention efforts. The few culturally specific cessation interventions that have been done have focused mostly on Mexicans in the Southwest and California1,2,3. Considering the diversity of the Latino population in the US, those interventions may not generalize to Latinos in the Northeast, who are mostly of Puerto Rican and Dominican origin. Research is limited in the area of HIV among Latinos and there are no studies to date that address the problem of tobacco use among HIV+ Latinos. We propose to address this disparity by focusing this particular research study on Latino men and women living with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Be receiving care for HIV at one of the participating immunology clinics
* Self-identify as being Latino/Hispanic (defined as being 1st, 2nd or 3rd generation from any of the Spanish-speaking countries of North America, Central America, South America and the Caribbean).
* Be 18 years old or older.
* Be current smokers of cigarettes (past 7 days)
* Speak English or Spanish

Exclusion Criteria:

* Are pregnant or nursing
* Have uncontrolled hypertension
* Use other forms of tobacco like cigars or chewing tobacco or are using anything else to help them quit smoking
* Are allergic to the nicotine patch or have a skin condition like eczema or psoriasis that makes them unable to use the patch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Stanton, Ph.D., Principal Investigator — Butler Hospital/Brown University
Locations (8):
- United States (8):
  - Lowell Community Health Center, Lowell, Massachusetts
  - Greater New Bedford Community Center, New Bedford, Massachusetts
  - Dimock Community Health Center, Roxbury, Massachusetts
  - Family Health Center of Worcester, Worcester, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Rhode Island Hospital HIV Clinic, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - The Miriam Hospital Immunology Clinic, Providence, Rhode Island

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506